CLINICAL TRIAL: NCT03057262
Title: The Efficiency of Anterior Repositioning Splint for the Management of Pain Related to Temporomandibular Joint Disc Displacement With Reduction
Brief Title: The Efficiency of Anterior Repositioning Splint for the Management of Temporomandibular Joint Dysunction
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Malgorzata Pihut, Associate Professor, Jagiellonian University
Other Study IDs: 122.6120.43.2016 BC
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Temporomandibular Joint Disc Displacement
Keywords: temporomandibular joint disorders; disc displacement with reduction; anterior repositioning splint
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Study group: Study group consisted of 56 subjects of both genders with unilateral or bilateral disc displacement(s) with reduction and pain in the area of temporomandibular joint. Patients were recruited from the Consulting Room of Temporomandibular Joint Dysfunction at the Jagiellonian University in Krakow during the years 2014-2016. In the study group was used the typical acrylic anterior repositioning splint fabricated in tete-a-tete (incisal) jaws position, covered the lower teeth arch to recapture a displaced disc(s) and decrease the intensity of pain. The anterior repositioning splint was recommended to 20 - hour use for a period of four months.
  Interventions: Device: Repositioning splint
- Control group: Control group consisted of 56 subjects of both genders with unilateral or bilateral disc displacement(s) with reduction and pain in the area of temporomandibular joint. Patients were recruited from the Consulting Room of Temporomandibular Joint Dysfunction at the Jagiellonian University in Krakow during the years 2014-2016. In the control group the investigators used the biostymulation laser (Terapus 2, Accuro, Poland), wave length 808 nm, power 32 J in the form of 12 session (duration of a single session was 3 min 45 s), performed every second day, on the area of the both temporomandibular joints (distance to the skin was 1 cm) with opened mouth and systematic performing of muscles self-exercises with a dominant protrusive position of mandible.

INTERVENTIONS:
Device: Repositioning splint — Application of repositioning splint in the study group.
  Groups: Study group

SUMMARY:
Intra-articular temporomandibular disorders are often related to pain in the area of temporomandibular joint, ear and temple. The aim of the study was to investigate the efficiency of anterior repositioning splints for the management of pain related to temporomandibular joint disc displacement with reduction.

DETAILED DESCRIPTION:
The research material consisted of 112 patients, aged 24 to 45 years, of both genders, who reported to the treatment in Consulting Room of Temporomandibular Joint Dysfunctions at the Jagiellonian University in Cracow, between 2014-2016, due to the pain and clicking of temporomandibular joints with comorbid hypertension of masticatory muscles. Subjects were examined according to the Diagnostic Criteria for Temporomandibular Disorders protocol and after inclusion with painful disc displacement with reduction and masticatory muscle contracture assigned randomly to the study or control group (56 patients in each). In the study group was used the anterior repositioning splint on the lower arch for 20 hour usage per 4 months. In the control group a non-invasive therapy was applied using biostimulation laser in the form of 12 session, performed every second day, on the area of the temporomandibular joints with opened mouth and performing muscles self-exercises with a dominant protrusive position of the mandible. Pain intensity was evaluated using verbal numerical rating scale (VNRS) immediately before the treatment and then after 4 and 16 weeks. The obtained data were analyzed using U Mann-Whitney test (p ≤ 0,005).

ELIGIBILITY:
Inclusion Criteria:

1. unilateral or bilateral presence of clicking, popping and/or snapping noise(s) detected with palpation during opening or closing or lateral or protrusive movements in TMJ(s),
2. in the previous 30 days, any TMJ noise(s) present with jaw movement or function,
3. unilateral or bilateral pain in the area of temporomandibular joint,
4. presence of masticatory muscles contracture,
5. full dentition or single tooth loss,
6. good general health,
7. positive mandible protrusion test,
8. no contraindications for laser therapy
9. patient consent to be involved in the study.

Exclusion Criteria:

1. partial tooth loss or edentulism,
2. contraindications for laser therapy
3. absence of appropriate symptoms
4. absence of consent to be involved in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 112 subjects were included to the study, 83 women and 29 men aged 24-45 years (mean age was 31). The study group includes 40 women and 16 men, and the control group contains 43 women and 13 men.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain relief related to temporomandibular joint disc displacement with reduction | 16 weeks
  Repositioning splint was applied to check its efficiency of pain relieving in a case of temporomandibular joint disc displacement with reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Pihut, DDS, PhD, Study Director — Jagiellonian University; Malgorzata Gorecka, DDS, Principal Investigator — Jagiellonian University; Piotr Ceranowicz, MD, PhD, Study Chair — Jagiellonian University; Mieszko Wieckiewicz, DMD, PhD, Study Chair — Wroclaw Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pihut M, Gorecka M, Ceranowicz P, Wieckiewicz M. The Efficiency of Anterior Repositioning Splints in the Management of Pain Related to Temporomandibular Joint Disc Displacement with Reduction. Pain Res Manag. 2018 Feb 21;2018:9089286. doi: 10.1155/2018/9089286. eCollection 2018. PMID 29682131